CLINICAL TRIAL: NCT05628831
Title: COMPARISON BETWEEN AUTOLOGOUS TISSUE RECONSTRUCTION USING vNOTES AND TRADITIONAL SURGERY IN TREATMENT OF PELVIC ORGAN PROLAPSE
Brief Title: Traditional Vaginal Surgery VS Autologous Tissue in Pelvic Floor Repair
Acronym: PREFAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital Zadar (Other)
Responsible Party: Principal Investigator, Luka Matak M.D., univ.mag spec Luka Matak M.D., General Hospital Zadar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GHZadar
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Vaginal Vault Prolapse
Keywords: Autologous graft; vNOTES; Pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: In one group of patients vaginal hysterectomy will be done with anterior and/or posterior repair depending on the judgment of the surgeon at the time of the operation. Second group will be treated with minimally invasive technique (vNOTES-vaginal natural orifice transluminal surgery) in which we will remove uterus and support pelvic floor with autologous tissue. Tissue graft will be isolated from abdominal rectus muscle. Fixation will be done using vNOTES aproach.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional surgery (Placebo Comparator): This group of patients will be treated with standard technique (vaginal hysterectomy with anterior and/or posterior vaginal repair) for pelvic organ prolapse .
  Interventions: Procedure: Vaginal surgery
- vNOTES PREFAP (Active Comparator): This group of patients will be treated with vNOTES aproach using autologous graft isolated from posterior rectus fascia for pelvic organ prolapse.
  Interventions: Procedure: vNOTES suspension with autologous tissue

INTERVENTIONS:
Procedure: vNOTES suspension with autologous tissue — Autologous tissue will be fixated on solid points in pelvis using vNOTES.
  Arms: vNOTES PREFAP
Procedure: Vaginal surgery — Vaginal hysterectomy will be done with anterior and/or posterior repair depending on the judgment of the surgeon at the time of the operation. Uterosacral and cardinal ligaments will be repositioned and attached to the vaginal vault after hysterectomy at the time of vault closure. A modified McCall culdoplasty will be done in this group to prevent enterocele and further apical prolapse
  Arms: Traditional surgery

SUMMARY:
The goal of this randomized, non blind, one center study is to compare the efficacy of vNOTES (vaginal natural orifice transluminal surgery) and traditional vaginal operation between the two groups by determining the risk of re-operation for anterior, posterior or apical prolapse within the study period.

Participants with a POP-Q (Pelvic Organ Prolapse Quantification) of 3 or 4 and an indication for hysterectomy and prolapse repair will be selected and randomly divided in two groups. One group will be operated with standard technique for pelvic organ prolapse and in the other autologous graft will be used using vNOTES ICIQ-LUTSqol (International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire IUGA revised (PISQ-IR) will be used as a subjective measurement of operative treatment.

Objective evaluation of the effect of postoperative results will be done using transperineal ultrasound before operation, 6 and 12 months after procedure.

EXPECTED CONTRIBUTION: In this research we will evaluate the feasibility and surgical outcome of vaginal NOTES (vNOTES) prolapse repair using posterior rectus fascia (PREFAP- Posterior Rectus Fascia Prolapse repair)

DETAILED DESCRIPTION:
All patients will be operated by the same surgeon. Antibiotic prophylaxis will be given pre-operatively according hospital protocols 30 minute before surgery. Surgery will be performed under general anesthesia in the lithotomy position with legs in stirrups The following peri-operative and patient data will be collected and analyzed: preoperative POP- Q, body mass index (BMI), age, parity, history of vaginal delivery, previous pelvic surgery, total operating time, estimated bloodloss, serum hemoglobin (Hb) drop (change between preoperative Hb and postoperative Hb 1 day after surgery), peri-operative complications, post- operative pain score and POP-Q after 6 and 12 months.

The ICIQ-LUTSqol questionnaire (International Consultation on Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module) is a psychometrically robust patient- completed questionnaire evaluating quality of life (QoL) in urinary incontinent patients with particular reference to social effects. It has 20 items to response with overall score between 19- 76 indicating increased impact on quality of life with greater values.

Subjective surgical outcome was measured using the Patient Global Impression of Improvement (PGI-I), which is a validated tool as a global index of response to prolapse surgery. The PGI-I is a seven-scale response for women comparing the postoperative condition with the pre-operative state, 1 being very much better and 7 being very much worse.

The women's prolapse symptoms and their impact will be evaluated before surgical treatment. A subjective assessment of the prolapse was made using Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire IUGA revised (PISQ-IR) before and 12 months after treatment. The PISQ-IR is designed as a condition-specific measure of sexual function in women with pelvic floor dysfunction, including urinary and anal incontinence and pelvic organ prolapse. It consists on 18-21 questions depending weather respondent indicates having a sexual partner or not. The cutoff score of 2.68 for PISQ-IR Summary Score allowed to diagnose sexual dysfunction in sexually active women with pelvic floor disorders.

Pelvic floor ultrasound will be performed before the operation and at 6 and 12 months after the operation. The inspection methods are as follows: Before the inspection, patients emptied the stool and moderately filled the bladder. The following parameters will be measured in resting state using the maximal Valsalva maneuver: Posterior vesicourethral angle (PVA):This included the angle between the proximal urethra and posterior wall of the bladder. Urethral tilt angle: This included the angle between the proximal urethra and vertical axis of the human body. Value is negative if the urethral axis deviated to the ventral side, and the value was positive when it is deviated to the dorsal side. Postoperative rotation angle of the urethra (UR): This refers to the difference in PVA between the Valsalva state and resting state. Bladder neck descent (BND): This refers to the vertical displacement of the bladder neck between the Valsalva state and resting state.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old with no desire to preserve fertility, POP-Q 3 or 4 stage of prolapse with indication for hysterectomy (abnormal uterine bleeding, enlarged fibrous uterus, premalignant cervical findings)

Exclusion Criteria:

* Virginity, pregnancy, acute urinary infection were considered contraindications; malignancy, previous PID or rectal surgery. Rectovaginal endometriosis. Contraindication for general anaesthesia, pneumoperitoneum or Trendelenburg position. Previous pelvic radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Traditional surgery vrs vNOTES PREFAP | 1 year
  Compare the efficacy of vNOTES autograft repair and traditional surgery between the two groups by determining the risk of reoperation for anterior, posterior or apical prolapse within the study period

SECONDARY OUTCOMES:
Complications | 1 year
  Diagnosis of an autologous tissue or vNOTES-associated complication.
QoL | 1 year
  Compare quality of life in both groups before operation and 6 months after procedure using ICIQ-LUTSqol questionnaire
Subjective pelvic floor outcomes | 1 year
  Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire IUGA revised (PISQ-IR) will be used before and 12 months after treatment to compare subjective impression of procedure
Ultrasound measurement | 1 year
  Objective evaluation of the effect of postoperative results using transperineal ultrasound before operation, 6 and 12 months after procedure
Learning curve | 1 year
  To assess the learning curve of harvesting the PREFAP autologous tissue measuring time and complications

CONTACTS AND LOCATIONS:
Locations (1):
- Luka Matak MD, Zadar, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All data relevant to the research results will be published
Supporting Information: Study Protocol
Time Frame: After the end of follow up period data will be available for one months

REFERENCES:
- [Result] Hokenstad ED, Glasgow AE, Habermann EB, Occhino JA. Readmission and Reoperation After Surgery for Pelvic Organ Prolapse. Female Pelvic Med Reconstr Surg. 2017 Mar/Apr;23(2):131-135. doi: 10.1097/SPV.0000000000000379. PMID 28067747
- [Result] Glazener CM, Breeman S, Elders A, Hemming C, Cooper KG, Freeman RM, Smith AR, Reid F, Hagen S, Montgomery I, Kilonzo M, Boyers D, McDonald A, McPherson G, MacLennan G, Norrie J; PROSPECT study group). Mesh, graft, or standard repair for women having primary transvaginal anterior or posterior compartment prolapse surgery: two parallel-group, multicentre, randomised, controlled trials (PROSPECT). Lancet. 2017 Jan 28;389(10067):381-392. doi: 10.1016/S0140-6736(16)31596-3. Epub 2016 Dec 21. PMID 28010989
- [Result] Seth J, Toia B, Ecclestone H, Pakzad M, Hamid R, Greenwell T, Ockrim J. The autologous rectus fascia sheath sacrocolpopexy and sacrohysteropexy, a mesh free alternative in patients with recurrent uterine and vault prolapse: A contemporary series and literature review. Urol Ann. 2019 Apr-Jun;11(2):193-197. doi: 10.4103/UA.UA_85_18. PMID 31040607
- [Result] Sharifiaghdas F. Autologous rectus fascia graft in the treatment of high-stage apical vaginal prolapse: preliminary results of a new surgical approach with native tissue. Int Urol Nephrol. 2022 May;54(5):1017-1022. doi: 10.1007/s11255-022-03167-8. Epub 2022 Mar 14. PMID 35286581
- [Result] Gon LM, Riccetto CLZ, Coltro Neto F, Achermann APP, Pereira TA, Palma PCR. Sacrospinous hysteropexy with an autologous rectus fascia sling for treatment of advanced apical pelvic organ prolapse. Int Urogynecol J. 2021 Aug;32(8):2291-2293. doi: 10.1007/s00192-021-04747-5. Epub 2021 Mar 17. PMID 33730231
- [Result] Lee JC, Olaitan OK, Lopez-Soler R, Renz JF, Millis JM, Gottlieb LJ. Expanding the envelope: the posterior rectus sheath-liver vascular composite allotransplant. Plast Reconstr Surg. 2013 Feb;131(2):209e-218e. doi: 10.1097/PRS.0b013e3182789c28. PMID 23358016
- [Result] Agarwal S, Dorafshar AH, Harland RC, Millis JM, Gottlieb LJ. Liver and vascularized posterior rectus sheath fascia composite tissue allotransplantation. Am J Transplant. 2010 Dec;10(12):2712-6. doi: 10.1111/j.1600-6143.2010.03331.x. PMID 21114648
- [Result] Ravindra KV, Martin AE, Vikraman DS, Brennan TV, Collins BH, Rege AS, Hollenbeck ST, Chinappa-Nagappa L, Eager K, Cousino D, Sudan DL. Use of vascularized posterior rectus sheath allograft in pediatric multivisceral transplantation--report of two cases. Am J Transplant. 2012 Aug;12(8):2242-6. doi: 10.1111/j.1600-6143.2012.04088.x. Epub 2012 May 17. PMID 22594310
- [Result] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BWJ, Bosteels JJA. Transvaginal natural orifice transluminal endoscopic surgery (vNOTES) adnexectomy for benign pathology compared with laparoscopic excision (NOTABLE): a protocol for a randomised controlled trial. BMJ Open. 2018 Jan 10;8(1):e018059. doi: 10.1136/bmjopen-2017-018059. PMID 29326183